CLINICAL TRIAL: NCT05457972
Title: Postpartum Vaginal Estrogen for Sexual Function in Breastfeeding Patients: A Randomized Controlled Trial
Brief Title: Postpartum Vaginal Estrogen for Breastfeeding Patients
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Rachel Pope, Clinical Instructor, Obstetrics and Gynecology - CWRU School of Medicine, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY20220578
Record Dates: First submitted 2022-07-11; First posted 2022-07-14 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-03

CONDITIONS: Breastfeeding; Postpartum Sexual Dysfunction; Vaginal Atrophy
Keywords: vaginal atrophy; postpartum; sexual dysfunction; dyspareunia; breastfeeding; pumping; vaginal dryness
MeSH Terms: conditions — Breast Feeding; Sexual Dysfunction, Physiological; Dyspareunia | interventions — Estradiol

STUDY DESIGN:
Intervention Model Description: Patients will be randomized in a 1:1 ratio into two study groups: vaginal estrogen or vaginal moisturizer. Randomization will be performed using blocking with a block size of 10 and a 1:1 allocation ratio. The randomization sequence will be generated using a random number table.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Vaginal Estrogen (Experimental): Estradiol 4 mcg vaginal insert, daily for two weeks then twice weekly for ten weeks.
  Interventions: Drug: Estradiol
- Vaginal Moisturizer (Active Comparator): Vaginal moisturizer, daily for two weeks then twice weekly for ten weeks.
  Interventions: Device: Vaginal Moisturizer

INTERVENTIONS:
Drug: Estradiol — Imvexxy is an FDA-approved drug produced by TherapeuticsMD.
  Other Names: Imvexxy
  Arms: Vaginal Estrogen
Device: Vaginal Moisturizer — Ingredients include hydrogenated coconut and palm oils and natural-source vitamin E (d-alpha tocopheryl acetate and tocopherols).
  Other Names: Carlson Key-E Suppositories
  Arms: Vaginal Moisturizer

SUMMARY:
Sexual dysfunction is very common in the postpartum period and is more common in people who breastfeed or pump. This research study was designed to help determine whether postpartum patients who use vaginal estrogen cream while breastfeeding have improved sexual function compared to postpartum patients who do not.

DETAILED DESCRIPTION:
This will be a prospective, randomized clinical trial of postpartum breastfeeding patients. Postpartum patients at University Hospitals (UH) MacDonald Women's Hospital will be evaluated for inclusion/exclusion by review of their medical record by the study investigators prior to discharge home. The study will then be discussed with the eligible patients privately. If they agree to participate, informed consent will be obtained. At this time, contact information will be obtained for all consenting patients.

Between 5 and 6 weeks postpartum, all consented patients will be contacted via their preferred form of communication. Inclusion criteria and desire for continued study participation will be verified prior to randomization. A baseline REDCap questionnaire will be texted or emailed to confirmed study participants. UH REDCap is a HIPAA-certified, secure, web-based data storage platform for research studies.

The patient will then be randomized in a 1:1 ratio into two study groups: vaginal estrogen or vaginal moisturizer. Randomization will be performed using blocking with a block size of 10 and a 1:1 allocation ratio. The randomization sequence will be generated using a random number table.

After randomization, but not prior to 6 weeks postpartum, the investigational drug service courier service will deliver softgel inserts of vaginal estrogen to the homes of participants randomized to the estrogen arm. Study investigators will deliver vaginal moisturizer to the homes of participants randomized to the placebo arm. Study participants will be provided with an instructional handout including information about how and how often to use the inserts or the moisturizer. Participants will be instructed to start using the inserts or lubricant when they receive the delivery. This will be considered the start of the study period.

During the study period, participants will use either estrogen or vaginal moisturizer nightly for two weeks and then twice weekly for ten weeks. Each week during the study period, participants will receive a message via their preferred communication method with five questions:

* Did you breastfeed or pump this week?
* Were you sexually active this week?
* If you were sexually active, did you have vaginal pain with sexual activity?
* How many times this week did you use the vaginal insert?
* Did you experience any change in your health this week?

  6 and 12 weeks into the study period, the patient will be contacted by their preferred communication method and requested to complete a questionnaire via UH REDCap.

The initial study questionnaire will include questions about demographics, gravidity and parity, prior deliveries (including mode of delivery, obstetric lacerations, and infant feeding), baseline sexual activity, prior pelvic surgery, chronic pain disorders, and plans for infant feeding. The 6 and 12-week study questionnaires will include the FSFI, the GAD-7 anxiety questionnaire, the Edinburgh Postnatal Depression Scale (EPDS), and the urinary distress inventory (UDI-6), the vaginal assessment scale (VAS), the Sexual Function Questionnaire Medical Impact Scale (SFQ-MIS), and the Female Sexual Distress Scale-Revised (FSDS-R) as well as questions about sexual activity and plans for infant feeding.

Questionnaire responses will be reviewed by a study investigator after completion by the patient. Any patients whose questionnaires indicate possible depression (EPDS score 10+), thoughts of self-harm (any answer other than "never" on EPDS question 10), or moderate to severe anxiety (GAD-7 score 10+) will be evaluated for safety by a physician study investigator and referred to UH Reproductive Behavioral Health.

In order to assess long term benefits of estrogen therapy in the early postpartum period, additional questionnaires will be administered at 6 months and 1 year to patients. The study intervention period will last 12 weeks, after which no additional vaginal estrogen or vaginal moisturizer will be administered to participants. Patients desiring to continue treatment after the 12-week study intervention period will be referred to their postpartum care provider. Patients will be instructed to stop estrogen use after they have completed breastfeeding.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Sexually active
* Singleton, term (37 weeks 0 days) birth
* Planning to breastfeed or pump during the study period
* History of successful breastfeeding or pumping after a prior pregnancy
* Between 6 weeks and 6 months postpartum (patients may be recruited at any time during the postpartum period, but the study period will not start until 6 weeks postpartum)
* Ability to consent in English
* Not meeting any exclusion criteria

Exclusion Criteria:

* Preterm delivery
* Perinatal mortality
* History of difficulty breastfeeding
* 3rd or 4th degree perineal laceration
* Any contraindications to estrogen, including, but not limited to, breast cancer or a history of breast cancer, estrogen-dependent neoplasia, active deep vein thrombosis (DVT)/pulmonary embolism (PE) or a history of these conditions, active arterial thromboembolic disease (for example, stroke and MI) or a history of these conditions, known anaphylactic reaction, angioedema, or hypersensitivity to estrogen, hepatic impairment or disease, protein C, protein S, or antithrombin deficiency, or other known thrombophilic disorders.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-02-22 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Total Female Sexual Function Index (FSFI) score | Up to 12 weeks into study period
  Female Sexual Function Index (FSFI) overall score has six domains and a maximum score of 36, with a higher score indicating better functioning. A score of 26 has been validated as a threshold for diagnosing female sexual dysfunction.

SECONDARY OUTCOMES:
Desire as measured by Female Sexual Function Index (FSFI) | Up to 12 weeks into study period
  One out of six FSFI domains. Score range of 1.2-6, with a higher score indicating better functioning.
Arousal as measured by Female Sexual Function Index (FSFI) | Up to 12 weeks into study period
  One out of six FSFI domains. Score range of 0-6, with a higher score indicating better functioning.
Lubrication as measured by Female Sexual Function Index (FSFI) | Up to 12 weeks into study period
  One out of six FSFI domains. Score range of 0-6, with a higher score indicating better functioning.
Orgasm as measured by Female Sexual Function Index (FSFI) | Up to 12 weeks into study period
  One out of six FSFI domains. Score range of 0-6, with a higher score indicating better functioning.
Satisfaction as measured by Female Sexual Function Index (FSFI) | Up to 12 weeks into study period
  One out of six FSFI domains. Score range of 0.8-6, with a higher score indicating better functioning.
Pain as measured by Female Sexual Function Index (FSFI) | Up to 12 weeks into study period
  One out of six FSFI domains. Score range of 0-6, with a higher score indicating better functioning.
Intercourse resumption | Up to 12 weeks into study period
  Number of weeks until resumption of intercourse after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Pope, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Agarwal SK, Kim J, Korst LM, Hughes CL. Application of the estrogen threshold hypothesis to the physiologic hypoestrogenemia of lactation. Breastfeed Med. 2015 Mar;10(2):77-83. doi: 10.1089/bfm.2014.0030. Epub 2015 Jan 7. PMID 25565323
- [Background] Banaei M, Moridi A, Dashti S. Sexual Dysfunction and its Associated Factors After Delivery: Longitudinal Study in Iranian Women. Mater Sociomed. 2018 Oct;30(3):198-203. doi: 10.5455/msm.2018.30.198-203. PMID 30515059
- [Background] Constantine GD, Simon JA, Pickar JH, Archer DF, Kushner H, Bernick B, Gasper G, Graham S, Mirkin S; REJOICE Study Group. The REJOICE trial: a phase 3 randomized, controlled trial evaluating the safety and efficacy of a novel vaginal estradiol soft-gel capsule for symptomatic vulvar and vaginal atrophy. Menopause. 2017 Apr;24(4):409-416. doi: 10.1097/GME.0000000000000786. PMID 27922936
- [Background] Kahan BC, Jairath V, Dore CJ, Morris TP. The risks and rewards of covariate adjustment in randomized trials: an assessment of 12 outcomes from 8 studies. Trials. 2014 Apr 23;15:139. doi: 10.1186/1745-6215-15-139. PMID 24755011
- [Background] Krause M, Wheeler TL 2nd, Richter HE, Snyder TE. Systemic effects of vaginally administered estrogen therapy: a review. Female Pelvic Med Reconstr Surg. 2010 May;16(3):188-95. doi: 10.1097/SPV.0b013e3181d7e86e. PMID 22453284
- [Background] Matthies LM, Wallwiener M, Sohn C, Reck C, Muller M, Wallwiener S. The influence of partnership quality and breastfeeding on postpartum female sexual function. Arch Gynecol Obstet. 2019 Jan;299(1):69-77. doi: 10.1007/s00404-018-4925-z. Epub 2018 Oct 16. PMID 30327862
- [Background] McCabe MP, Sharlip ID, Lewis R, Atalla E, Balon R, Fisher AD, Laumann E, Lee SW, Segraves RT. Incidence and Prevalence of Sexual Dysfunction in Women and Men: A Consensus Statement from the Fourth International Consultation on Sexual Medicine 2015. J Sex Med. 2016 Feb;13(2):144-52. doi: 10.1016/j.jsxm.2015.12.034. PMID 26953829
- [Background] Portman DJ, Gass ML; Vulvovaginal Atrophy Terminology Consensus Conference Panel. Genitourinary syndrome of menopause: new terminology for vulvovaginal atrophy from the International Society for the Study of Women's Sexual Health and the North American Menopause Society. Menopause. 2014 Oct;21(10):1063-8. doi: 10.1097/GME.0000000000000329. PMID 25160739
- [Background] Shifren JL, Monz BU, Russo PA, Segreti A, Johannes CB. Sexual problems and distress in United States women: prevalence and correlates. Obstet Gynecol. 2008 Nov;112(5):970-8. doi: 10.1097/AOG.0b013e3181898cdb. PMID 18978095
- [Background] Suckling J, Lethaby A, Kennedy R. Local oestrogen for vaginal atrophy in postmenopausal women. Cochrane Database Syst Rev. 2006 Oct 18;(4):CD001500. doi: 10.1002/14651858.CD001500.pub2. PMID 17054136
- [Background] Alp Yilmaz F, Sener Taplak A, Polat S. Breastfeeding and Sexual Activity and Sexual Quality in Postpartum Women. Breastfeed Med. 2019 Oct;14(8):587-591. doi: 10.1089/bfm.2018.0249. Epub 2019 Jul 12. PMID 31298557